CLINICAL TRIAL: NCT02430805
Title: Genetics and Genomics of Hypertension Associated With Microinflammation, Oxydative Stress, Chronic Renal Disease and Heart Failure (A2-B2-B3)
Brief Title: Predisposition and Transition Mechanisms From Arterial Hypertension to Heart Failure
Acronym: Hypercare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Network of Excellence 6 PCRD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HYPERCARE(english v. 1.0)JRPB3; Cpp : 07.11.11; Dgs: 2007-0537
Record Dates: First submitted 2010-02-05; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2010-02

CONDITIONS: Hypertension
Keywords: hypertension; microinflammation and oxidative stress; renal disease; heart failure; genetics markers; genomics markers; proteomics markers
MeSH Terms: conditions — Hypertension; Kidney Diseases; Heart Failure | interventions — Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NOE (Other): multicentric family-based cohort. prospective and transversal study
  Interventions: Other: dna extraction and genotyping

INTERVENTIONS:
Other: dna extraction and genotyping — blood and urine sample

SUMMARY:
This project aims at investigating the genetic, genomic and proteomic basis of hypertension and susceptibility to hypertension-related end organ damage (renal damage and heart failure). It will include cross sectional as well as follow-up studies with a large number of subjects and variety of phenotypes, to explore the pathophysiology of hypertension and hypertension-related disease.

DETAILED DESCRIPTION:
In all index patients and recruited family members, recorded data will include the following :

* Past medical history, drug history and family history
* Physical examination
* Height, weight, waist and hip circumference
* Cardiac examination
* Vascular examination
* Blood pressure
* Plasma and urine samples
* Body composition (DEXA)
* Tissue Doppler imaging

ELIGIBILITY:
Inclusion Criteria:

* index patient :

  * Caucasian patients of either sex who were diagnosed to have essential hypertension (as defined below) before the age of 50 y.
  * The index patient should not be older than 60 years at the time of enrolment.
  * Definition of hypertension for the index patient:

    * If untreated: Systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 95 mmHg.
    * If already on treatment: Treatment with more of 2 different antihypertensive drugs at the time of enrolment.
  * At least three first degree relatives of whom at least one should be affected and at least one be from a different generation (parents or offspring aged 18 years or above) must be willing to participate in the family study. For definition of hypertension in relatives of the index patient see below.
  * Written informed consent
* family

  * at least three other first degree relatives must be willing to participate in the family study:
  * at least one first-degree relative must be affected with diagnosis of hypertension made before age of 50 years AND
  * at least one first degree relative must be from a different generation (offspring or parents).

Exclusion Criteria:

* index patient :

  * Any known form of secondary hypertension, including sleep apnoea syndrome
  * Any known previous clinical complications of hypertension (angina, MI, stroke, TIA, peripheral artery disease) at any time
  * Any known renal disease, including GFR < 60 mL/min as estimated by the abbreviated MDRD formula, or kidney stones
  * Kidney or other organ transplantation
  * Type 1 diabetes mellitus
  * Heart failure stage D (AHA/ACC criteria)
  * Any malignant concomitant diseases or history of malignant diseases within the last five years, with exception of treated squamous skin cancer or basalioma
  * Clinical or laboratory signs of acute infection, especially urinary tract infection
  * Systemic inflammatory diseases, such as autoimmune diseases, connective tissue diseases or collagenoses.
  * Steroids or any other immunosuppressive drug
  * Severe known liver disease (ALT or gamma-GT above three-fold of upper normal limit)
  * Current alcohol consume of more than 21 drinks/week (1 drink = a bottle (0,33 l) beer, a glass (0,2 l) of wine, or 4 cl = 40 ml of spirit (40%)) or drug abuse such as cocaine
* family

  * any organ transplantation
  * any malignant concomitant disease
  * acute infection
  * systemic inflammatory disease
  * severe liver disease
  * current alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
genetic biomarkers | time point 1 : first day ; Time point

SECONDARY OUTCOMES:
oxidative stress markers | time point 1 : first day ; Time point 2 : 2 years ; Time point 3 : 4 years
microinflammation markers | time point 1 : first day ; Time point 2 : 2 years ; Time point 3 : 4 years
renal function and damage markers | time point 1 : first day ; Time point 2 : 2 years ; Time point 3 : 4 years
cardiac and large artery growth, remodelling dysfunction and failure markers | time point 1 : first day ; Time point 2 : 2 years ; Time point 3 : 4 years

CONTACTS AND LOCATIONS:
Overall Officials: faiez ZANNAD, Pr, Principal Investigator — Central Hospital, Nancy, France
Locations (2):
- France (2):
  - Centre D'Investigation Clinique de Strasbourg, Strasbourg, Alsace
  - Hopital Brabois adulte, Nancy, Lorraine

REFERENCES:
- [Derived] Mandry D, Girerd N, Lamiral Z, Huttin O, Filippetti L, Micard E, Beaumont M, Ncho Mottoh MB, Pace N, Zannad F, Rossignol P, Marie PY. Relationship Between Left Ventricular Ejection Fraction Variation and Systemic Vascular Resistance: A Prospective Cardiovascular Magnetic Resonance Study. Front Cardiovasc Med. 2021 Dec 24;8:803567. doi: 10.3389/fcvm.2021.803567. eCollection 2021. PMID 35004914